CLINICAL TRIAL: NCT06976762
Title: Near-Infrared Spectroscopy Measurements in Patients With Chronic Obstructive Pulmonary Disease, and Chronic Renal Disease: An Observational Study
Brief Title: Near-Infrared Spectroscopy Measurements in Chronic Obstructive Pulmonary Disease
Acronym: NIRS
Status: Enrolling by invitation | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Serkan Dogru, Associate Professor, Tokat Gaziosmanpasa University
Other Study IDs: 20-KAEK-212
Record Dates: First submitted 2024-12-07; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Microcirculatory Status; Spectroscopic Analysis; COPD; Renal Failure
Keywords: microcirculation; spectroscopy; pulmonary disease; renal failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Renal Insufficiency; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD: Patients with aged between 18 and 80 years, a confirmed diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria, a post-bronchodilator forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) ratio of <0.70, and clinically stable COPD, with no exacerbations or hospital admissions within the preceding four weeks were enrolled in this COPD group.
- CKD: Patients with aged between 18 and 80 years, evidence of CKD, an estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73 m² (Stages 3-5 CKD) on at least two occasions three months apart, or a history of renal replacement therapy were enrolled in CKD group.
- Control: Healthy individuals

SUMMARY:
Participants were selected based on three groups: healthy, chronic obstructive pulmonary disease, and chronic renal disease. NIRS was used to measure tissue oxygenation on the thenar region of the right hand. A pressure cuff was used to temporarily occlude arterial inflow, thus allowing the response to this to be assessed. The StO2 was plotted against time, and the following variables were calculated, the downslope, upslope, area under curve.

DETAILED DESCRIPTION:
This study was a prospective observational analysis involving patients with diagnosed Chronic Obstructive Pulmonary Disease (COPD) and Chronic Kidney Disease (CKD). Participants were recruited from the pulmonary and nephrology clinics at Gaziosmanpasa University Health Application and Research Centre during their stay in the ward. The study was approved by the Tokat Gaziosmanpasa Research Ethics Committee (Grant number: 20-KAEK-212) and all patients provided informed consent prior to participation.

Data collection involved baseline assessments of demographic characteristics, COPD severity, renal function, and comorbidities. Participants were divided into three groups: control, COPD, and CRD. Patients were visited during their stay in the ward and the measurement was initiated after five minutes of rest. Venous blood gas analysis was performed using the same sample of blood obtained for routine complete blood count analysis. A vascular occlusion test was conducted with NIRS measurements taken throughout. Three minutes of baseline measurement placing the probe on thenar eminence of the right hand was completed while the patient was lying with 45 degrees back up position. After baseline measurements a non-invasive blood pressure cuff was placed on the right arm and it was inflated to 250 mmHg. The cuff was held inflated for two minutes; after two minutes, the cuff was deflated and the measurement had been continued for another three minutes and stopped. Near-infrared spectroscopy measurements were obtained during and after vascular occlusion, including the area under curve (AUC) during occlusion (representing tissue hyperemia) and the angles of descent and ascent, which reflect muscle oxygen consumption and microcirculatory function, respectively.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients were required to meet all of the following criteria:

  1. Age: Patients aged between 18 and 80 years.
  2. COPD Diagnosis: A confirmed diagnosis of COPD according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria, including:

     * A post-bronchodilator forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) ratio of <0.70.
  3. Renal Failure: Evidence of CKD, defined as:

     * An estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73 m² (Stages 3-5 CKD) on at least two occasions three months apart, or a history of renal replacement therapy.
  4. Stable Medical Condition: Clinically stable COPD, with no exacerbations or hospital admissions within the preceding four weeks.

Exclusion Criteria:

* Patients were excluded from the study if they met any of the following criteria:

  1. Acute Exacerbation: Evidence of an acute COPD exacerbation within four weeks prior to enrolment.
  2. Other Respiratory Disorders: Coexistence of other chronic respiratory diseases such as asthma, interstitial lung disease, or bronchiectasis that might interfere with the assessment of COPD.
  3. Renal Transplantation: History of kidney transplantation, as immunosuppressive therapy may affect disease progression and outcomes.
  4. Uncontrolled Comorbidities: Presence of any uncontrolled comorbid conditions, including:

     * Cardiovascular instability or recent myocardial infarction (within six months).
     * Active malignancy (other than localized skin cancer).
     * Severe liver disease (e.g., cirrhosis with hepatic failure).
  5. Pregnancy or Breastfeeding: Women who were pregnant or breastfeeding at the time of study enrolment.
  6. Cognitive Impairment: Any condition that would impair the ability to provide informed consent or participate in study procedures, such as dementia or significant psychiatric disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lipcsey et al.7 reported that the mean stO2 in volunteers was 80±7%.1 Based on this finding, assuming a 5% decrease in stO2 with a two-sided type I error of 0.05, and a power of 0.80; a total of 144 patients (each group consisted of 48 subjects) were required to find a significant difference between control, patients with COPD and patients with CRD groups.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
NIRS value-descent curve | two minutes
  After baseline measurements a non-invasive blood pressure cuff was placed on the right arm and it was inflated to 250 mmHg. The cuff was held inflated for two minutes; after two minutes, the cuff was deflated and the measurement had been continued for another three minutes and stopped. Near-infrared spectroscopy measurements were obtained during and after vascular occlusion, including the area under curve (AUC) during occlusion (representing tissue hyperemia) and the angles of descent and ascent, which reflect muscle oxygen consumption and microcirculatory function, respectively.
NIRS value-ascent curve | two minutes
  After baseline measurements a non-invasive blood pressure cuff was placed on the right arm and it was inflated to 250 mmHg. The cuff was held inflated for two minutes; after two minutes, the cuff was deflated and the measurement had been continued for another three minutes and stopped. Near-infrared spectroscopy measurements were obtained during and after vascular occlusion, including the area under curve (AUC) during occlusion (representing tissue hyperemia) and the angles of descent and ascent, which reflect muscle oxygen consumption and microcirculatory function, respectively.
NIRS value-area under curve | three minutes
  After baseline measurements a non-invasive blood pressure cuff was placed on the right arm and it was inflated to 250 mmHg. The cuff was held inflated for two minutes; after two minutes, the cuff was deflated and the measurement had been continued for another three minutes and stopped. Near-infrared spectroscopy measurements were obtained during and after vascular occlusion, including the area under curve (AUC) during occlusion (representing tissue hyperemia) and the angles of descent and ascent, which reflect muscle oxygen consumption and microcirculatory function, respectively.
NIRS value-baseline | three minutes
  After baseline measurements a non-invasive blood pressure cuff was placed on the right arm and it was inflated to 250 mmHg. The cuff was held inflated for two minutes; after two minutes, the cuff was deflated and the measurement had been continued for another three minutes and stopped. Near-infrared spectroscopy measurements were obtained during and after vascular occlusion, including the area under curve (AUC) during occlusion (representing tissue hyperemia) and the angles of descent and ascent, which reflect muscle oxygen consumption and microcirculatory function, respectively.

SECONDARY OUTCOMES:
blood gas analysis | one minute
  Venous blood gas analysis was performed using the same sample of blood obtained for routine complete blood count analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel MARTIN, Professor, Principal Investigator — Uni of Plymouth, Dept of Periop and ICU, Plymouth, UK
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It can be illegal to share the personal information of the individuals recruited in the study.